CLINICAL TRIAL: NCT00853034
Title: Effects of Arabinoxylan-Oligosaccharides on Colonic Metabolism and Microbial Composition Compared to Other Prebiotics in Healthy Subjects
Brief Title: Effects of Arabinoxylan-Oligosaccharides Compared to Other Prebiotics in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AXOS 001
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: gastrointestinal effects; prebiotic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOS-IN (Active Comparator): prebiotic fructo-oligosaccharide enriched inulin
  Interventions: Dietary Supplement: FOS-IN
- AXOS (Experimental): arabinoxylan-oligosaccharides (AXOS)
  Interventions: Dietary Supplement: AXOS

INTERVENTIONS:
Dietary Supplement: FOS-IN — prebiotic fructo-oligosaccharide enriched inulin
  intake period: 2 weeks, 1.25 or 2.50g every morning and evening
  Other Names: Synergy1, Orafti, Tienen
  Arms: FOS-IN
Dietary Supplement: AXOS — arabinoxylan-oligosaccharides (AXOS)
  intake period: 2 weeks, 1.25 or 2.50g every morning and evening
  Arms: AXOS

SUMMARY:
The purpose of the study is to evaluate the effects of arabinoxylan-oligosaccharides (AXOS) on the colonic metabolism and microbial composition, and to compare these effects with the reference prebiotic fructo-oligosaccharide enriched inulin.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* 18-45 years
* regular eating pattern

Exclusion Criteria:

* gastrointestinal complaints
* antibiotic intake
* medication influencing gut transit or microbiota
* abdominal surgery
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, PhD, Study Director — KU Leuven
Locations (1):
- Department of Gastrointestinal Research, Laboratory Digestion and Absorption, Leuven, Leuven, Belgium

REFERENCES:
- [Background] Cloetens L, De Preter V, Swennen K, Broekaert WF, Courtin CM, Delcour JA, Rutgeerts P, Verbeke K. Dose-response effect of arabinoxylooligosaccharides on gastrointestinal motility and on colonic bacterial metabolism in healthy volunteers. J Am Coll Nutr. 2008 Aug;27(4):512-8. doi: 10.1080/07315724.2008.10719733. PMID 18978172